CLINICAL TRIAL: NCT04702321
Title: Genetic Risks for Childhood Cancer Complications in Switzerland
Acronym: GECCOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Ansari, Professor Marc Ansari, University Hospital, Geneva
Other Study IDs: GECCOS
Record Dates: First submitted 2020-12-21; First posted 2021-01-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Childhood Cancer; Genetic Predisposition; Late Effect
Keywords: Childhood cancer; Late effects; Therapy complications; Second neoplasm; Registry; Biobank; Genetic variation; Genetic polymorphism; Pharmacogenetics; Genetic association studies
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Description: saliva, buccal swabs, blood, or other sample adequate for germline DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient cohort: Patients with clinical data and biospecimens
  Interventions: Other: Procedure: Biospecimen Collection; Other: Procedure: Medical Chart Review

INTERVENTIONS:
Other: Procedure: Biospecimen Collection — Collection of saliva, buccal swabs, blood, or other sample adequate for germline DNA extraction
  Other Names: Medical Chart Review
Other: Procedure: Medical Chart Review — Collection of clinical data
  Other Names: Registry data collection

SUMMARY:
The objectives of the GECCOS project are to identify genetic variants associated with complications of childhood cancer using genotype-phenotype association studies. Germline genetic samples and data of the "Germline DNA Biobank for Childhood Cancer and Blood Disorders Switzerland" (BISKIDS) which is included in the Geneva Biobank for Hematology and Oncology in Pediatrics (BaHOP) will be used with clinical data of Swiss childhood cancer patients collected at the Institute of Social and Preventive Medicine in Bern.

DETAILED DESCRIPTION:
Background and rationale :

Around 300 children and adolescents are diagnosed with cancer each year in Switzerland. A wide range of acute and chronic complications have been linked to cancer and its treatments. Cancer treatments, though highly curative, have a high incidence of adverse events, not only acutely but also chronically. Depending on the type and dose of treatments, the complications vary. There are important inter-individual differences in the type and severity of complications associated with similar cancer treatments. Genetic variation was identified to affect some complications and is suspected to play an important role in many of these differences.

The GECCOS project on analysis of genetic risks for complications associated with childhood cancers fills the gap to analyze germline genetic data with clinical information on short- and long-term complications. This has not been done on a nationwide scale in Switzerland yet. The GECCOS project will improve knowledge on germline genetic risks for complications and further personalize care during acute treatment and follow-up of childhood cancer patients.

Objectives:

Primary objectives:

1. Identify genetic variants associated with complications after childhood cancer leading to specific organ dysfunctions and second primary neoplasms.
2. Evaluate the functional importance of genetic variants for complications after childhood cancer through in silico and in vitro studies.

Secondary objective:

Assess genetic variants and their impact on multiple outcomes as a result of specific treatment exposures.

ELIGIBILITY:
Inclusion Criteria:

1. Registered in the Swiss Childhood Cancer Registry (SCCR) since 1976; AND
2. consented to the BaHOP (host biobank for the BISKIDS Biobanking project); AND
3. diagnosed with cancer according to the International Classification of Childhood Cancer, version 3, ICCC-3, or Langerhans cell histiocytosis (LCH) before age 21 years.

Exclusion Criteria:

1. Lacking written consent signed by participant and/ or their legal representative to participate in the BaHOP (where applicable); OR
2. died after study participation and declined use of their samples and data after their death in the original consent for BaHOP (as indicated on the BaHOP consent).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Brief description of the anticipated study population:
  Swiss childhood cancer patients and survivors are being invited to participate in the BaHOP biobank hosting the Germline DNA Biobank for Childhood Cancer and Blood Disorders Switzerland (BISKIDS). Recruitment for BISKIDS is done by the collaborators at the Institute of Social and Preventive Medicine (ISPM), University of Bern. As of December 2019, 9,306 persons were alive and eligible to participate in this project. Participants are invited in batches depending on inclusion criteria of specific sub-projects. Clinical data is collected at the ISPM for childhood cancer patients and survivors since 1976 which will be available for the GECCOS project for genotype-phenotype analysis.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic variants in participants as a possible marker of risk of complications after childhood cancer | Genetic sequencing performed at enrollment into study
  Genotyping of germline genetic variants (candidate gene, whole exome, or whole genome sequencing data)

SECONDARY OUTCOMES:
Number of participants with complications of childhood cancers: specific organ dysfunctions assessed by objective measurements and second primary neoplasms, extracted from medical records and cancer registry information | Data collection at enrollment into study, and longitudinal data collection until last follow-up or death from any cause, approx. 10 years
  * Specific organ dysfunctions assessed by objective measurements, e.g. audiograms for hearing loss, and self-assessment with questionnaires and
  * Second primary neoplasms as defined by the International Agency for Research on Cancer (IARC) criteria
Demographic and clinical covariates corresponding to possible risk factors for specific complications after childhood cancer, extracted from medical records and cancer registry information | Data collection at enrollment into study, and longitudinal data collection until last follow-up or death from any cause, approx. 10 years
  Covariates include but are not restricted to the collection of the following data:
  * demographic information, e.g. sex, age and year at diagnosis, etc.
  * cancer-related information, e.g. cancer type, stage, metastases, etc.
  * treatment-related risk factors, e.g. platinum chemotherapy exposure (with cumulative dose, mg/m2) for hearing impairment, radiation dose (gray) and fields for radiation toxicity, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Upon specific request to study PI (Marc.Ansari@hcuge.ch or: biskids@cansearch.ch)

REFERENCES:
- [Derived] Waespe N, Strebel S, Nava T, Uppugunduri CRS, Marino D, Mattiello V, Otth M, Gumy-Pause F, Von Bueren AO, Baleydier F, Mader L, Spoerri A, Kuehni CE, Ansari M. Cohort-based association study of germline genetic variants with acute and chronic health complications of childhood cancer and its treatment: Genetic Risks for Childhood Cancer Complications Switzerland (GECCOS) study protocol. BMJ Open. 2022 Jan 24;12(1):e052131. doi: 10.1136/bmjopen-2021-052131. PMID 35074812
- [Derived] Waespe N, Strebel S, Marino D, Mattiello V, Muet F, Nava T, Schindera C, Belle FN, Mader L, Spoerri A, Kuehni CE, Ansari M. Predictors for participation in DNA self-sampling of childhood cancer survivors in Switzerland. BMC Med Res Methodol. 2021 Oct 30;21(1):236. doi: 10.1186/s12874-021-01428-1. PMID 34717553